CLINICAL TRIAL: NCT05834374
Title: Training for Transfer by Contextual Variation: A Randomized Study
Brief Title: Training for Transfer by Contextual Variation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vilma Johnsson, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H-19039518
Record Dates: First submitted 2023-04-03; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Medical Education
Keywords: Medical education; Affordances; Contextual variation; Invasisve ultrasound skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Contextual variation (Experimental): The contextual variation group alternate between six affordance conditions where the surface of the model i either half covered combined with no guide, a partial guide or a complete guide.
  Interventions: Other: Contextual variation
- Maximum affordances (Experimental): The maximum affordances group has half the surface model covered and a complete guide throughout the session.
  Interventions: Other: Maximum affordances
- Minimum affordances (No Intervention): The control group has the whole surface uncovered and no guide throughout the session.

INTERVENTIONS:
Other: Contextual variation — The participants are instructed to perform ultrasound guided needle puncture of the cavities using a 20 ml syringe and a 15 cm, 18 Gauge biopsy needle. When all the three cavities are emptied the participant receive a new cube with refilled balloons. The new cube is equivalent to the old apart from being rotated 180 degrees. The participant are given one hour to empty as many cavities as possible. They are encouraged to track the needle with ultrasound while in the cube. The transfer test is performed on a CVS mannikin. The GE HealthCare LOGIQTM e Ultrasound is used with a C1-5 RS probe with or without the GE HealthCare C1-5 non-sterile ultrasound needle guide for both the training session and the transfer tests.
  Other Names: Maximum affordances
  Arms: Contextual variation
Other: Maximum affordances — The participants are instructed to perform ultrasound guided needle puncture of the cavities using a 20 ml syringe and a 15 cm, 18 Gauge biopsy needle. When all the three cavities are emptied the participant receive a new cube with refilled balloons. The new cube is equivalent to the old apart from being rotated 180 degrees. The participant are given one hour to empty as many cavities as possible. They are encouraged to track the needle with ultrasound while in the cube. The transfer test is performed on a CVS mannikin. The GE HealthCare LOGIQTM e Ultrasound is used with a C1-5 RS probe with or without the GE HealthCare C1-5 non-sterile ultrasound needle guide for both the training session and the transfer tests.
  Arms: Maximum affordances

SUMMARY:
The goal of this randomized study is to investigate the effect of introducing contextual variation on transfer when learning a technical skill in a group of medical students. The main questions it aims to answer is: If context variation of specific affordance conditions enhance the learner's ability to transfer out? Participants will practice performing an invasive ultrasound guided procedure either on a fantom with maximum affordances or with contextual variation. Researchers will compare the maximum affordances group and the contextual variation group to see if its effects compared to the control group with minimal affordances.

DETAILED DESCRIPTION:
Participants:

Participants are medical student from the University of Copenhagen. They are recruited by announcements on student fora on Facebook.

Randomization:

The participants are randomized to the intervention group contextual variation, the intervention group maximum affordances or control group minimum affordances in an 1:1:1 allocation ratio. In addition, the order of the four transfer tests (a, b, c and d) is randomly selected for each participant. The randomization was conducted by an independent research assistant at CAMES. Random permuted blocks are generated online for both the intervention and the transfer test.

Equiptment:

The training session is conducted on a ballistic gel cube. Three cavities are excavated corresponding to the points of a triangle at the bottom of the cube. Each cavity include a 5" latex balloon filled with 10ml water. The ballistic gel is coloured with graphite thus, the cavities can only be visualized by ultrasound. The participants are instructed to perform ultrasound guided needle puncture of the cavities using a 20 ml syringe and a 15 cm, 18 Gauge biopsy needle. When all the three cavities are emptied the participant receive a new cube with refilled balloons. The new cube is equivalent to the old apart from being rotated 180 degrees. The participant are given one hour to empty as many cavities as possible. They are encouraged to track the needle with ultrasound while in the cube. The transfer test is performed on a CVS mannikin. The GE HealthCare LOGIQTM e Ultrasound is used with a C1-5 RS probe with or without the GE HealthCare C1-5 non-sterile ultrasound needle guide for both the training session and the transfer tests.

Intervention:

In the first learning session the participants are provided with an ultrasound probe and a needle and instructed to detect and aim at a fixed target in a cube made of ballistic gel. The contextual variation group alternate between six affordance conditions where the surface of the model i either half covered combined with no guide, a partial guide or a complete guide. The maximum affordances group has half the surface model covered and a complete guide throughout the session. The control group has the whole surface uncovered and no guide throughout the session. The participants will have 60 minutes to complete the training.

Transfer test:

The groups are re-invited seven days after completed training for a transfer test. The transfer test include four cases (a, b, c, d) where the overall aim is to perform a CVS procedure on a CVS mannikin. In case a and b, the participant has the affordances of a guide on the ultrasound probe and the screen. In case c and d, there is a lack of affordances by not using a guide on the probe or screen. The placental position is anterior in case a and c, and posterior in case b and d. The transfer test measures both the transfer out, i.e. applying a skill learned in one context to a new context, and transfer in, how the learner learns with the acquired skills in the new context. The order of the transfer tests is randomized at inclusion. The participants receive a brief introduction to the chorionic villus sampling (CVS) procedure ahead of the transfer test by watching a video where the procedure is performed in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Passed a general anatomy exam
* Proficiency in Danish

Exclusion Criteria:

* Previous ultrasound experience except mandatory training as part of the medical curriculum

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Transfertest score | 4*7 min (4 tests) 7-10 days after intervention
  Exåpert based performances scores using a 5 point likert scale rating 4 items. Higher scores indicate better performance.

SECONDARY OUTCOMES:
Training | 60 min (training session)
  Quantitative analysis of use of movements (many movements indicate expert performance), number of emptied ballons (higher number indicates better perfomance), incisions/ballon (lower number indicates better performance)

CONTACTS AND LOCATIONS:
Overall Officials: Martin G Tolsgaard, Professor, Study Chair — Rigshospitalet, Denmark; Vilma L Johnsson, M.D., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Copenhagen Academy of Medical Education and Simulation, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Data can be shared upon request. However, raw data includes non-anonymized video records that are incompatible with sharing.